CLINICAL TRIAL: NCT03851172
Title: Nepafenac Versus Ketorolac Eye Drops in Prevention of Intraoperative Miosis During Cataract Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Mahrous Sayed, Resident at ophthalmology department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0925-0586
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cataract; Miosis
Keywords: Cataract surgery; Intraoperative Miosis; Ketorolac eye drops; Nepafenac eye drops
MeSH Terms: conditions — Cataract; Miosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Allocation concealment will be achieved by masking the bottles of the different agents which will be used in the study. All agents will be added to non-labeled bottles, then they will be labeled by the supervisor (who will not participate in eye drops administration) as bottle (1), bottle (2) and bottle (3). The most junior researcher will be responsible for the eye drops administration, for whom the different agents are not known.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nepafenac and cyclopentolate (Experimental): Nepafenac 1 mg eye drops two times before surgery and cyclopentolate eye drops two times before cataract surgery
  Interventions: Drug: Nepafenac Ophthalmic; Drug: Cyclopentolate Ophthalmic
- Ketorolac and cyclopentolate (Experimental): Ketorolac 0.5% eye drops two times before surgery and cyclopentolate eye drops two times before cataract surgery
  Interventions: Drug: Ketorolac Ophthalmic; Drug: Cyclopentolate Ophthalmic
- Cyclopentolate and saline 0.9% (Placebo Comparator): Cyclopentolate eye drops two times before surgery and saline 0.9% eye drops two times before cataract surgery
  Interventions: Drug: Cyclopentolate Ophthalmic

INTERVENTIONS:
Drug: Ketorolac Ophthalmic — Preoperative administration of Ketorolac 0.5% eye drops
  Arms: Ketorolac and cyclopentolate
Drug: Nepafenac Ophthalmic — Preoperative administration of Nepafenac 1 mg eye drops
  Arms: Nepafenac and cyclopentolate
Drug: Cyclopentolate Ophthalmic — Preoperative administration of Cyclopentolate eye drops

SUMMARY:
This study aim at determining the efficacy of Nepafenac and Ketorolac in obtaining adequate intraoperative mydriasis and preventing miosis during cataract surgery. It also compare the efficacy of both Nepafenac versus Ketorolac, and determine the more effective agent in preventing miosis during cataract surgery. The investigators try to determine if the effect of preoperative NSAIDs agents use would show a financial benefit, or this manoeuvre would add a financial load on the patients who are candidate for cataract surgery.

DETAILED DESCRIPTION:
Maintaining adequate mydriasis is one of the most important prerequisites during both extracapsular cataract extraction and phacoemulsification intervention. The importance of intraoperative maintenance of mydriasis arises from the necessity for the surgeon to insert intra-ocular lens in the posterior chamber of the eye. It is now well established that non-steroidal anti-inflammatory drugs (NSAIDs) reduce intraoperative miosis during cataract surgery. Topical Flurbiprofen, Indomethacin and Diclofenac with and without intraoperative epinephrine are the commonest topical non-steroidal eye drops with which nearly all publications in the literature studied the prevention of intraoperative surgery-induced miosis. In addition, Diclofenac was found to be the most effective NSAIDs agent in maintaining intraoperative mydriasis.

More recently, evidence that some NSAIDs, namely ketorolac and Flurbiprofen, may have a role in preventing pseudophakic cystoid macular oedema.

Patients whom eyes are pre-treated with some NSAIDs, especially diclofenac, shows a statistically significant reduction in the degree of postoperative inflammation (e.g., redness, pain and itching) on the first post-operative day. On the contrary, Thaller et al found, in his study at 2000, that no statistically significant difference in the postoperative redness, pain and cells in the anterior chamber.

Administration of Adrenalin in the anterior chamber fluid is found by several studies to be more effective in maintaining intraoperative mydriasis than preoperative treatment with NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract who are candidate for cataract surgery

Exclusion Criteria:

* D.M,
* Patient with other ocular comorbidities rather than cataract,
* Patients with history of trauma.
* Patients on Corticosteroid drops treatment.
* Previous intraocular surgery.

Ages: 2 Days to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of miosis during cataract surgery | 30 minutes
  The prevention of intraoperative miosis during cataract surgery after preparation by the different eye drops and cyclopentolate